CLINICAL TRIAL: NCT06881485
Title: Naltrexone/Bupropion With or Without Very Low Calorie Ketogenic Diet for Weight Regain After Bariatric Surgery
Acronym: Relay
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S68952
Record Dates: First submitted 2025-02-27; First posted 2025-03-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Weight Regain Post Bariatric Surgery; Obesity (Disorder)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexon/Bupropion + Lifestyle + VLCKD (Experimental): Naltrexon/Bupropion + Lifestyle + VLCKD
  Interventions: Other: Very Low Calorie Diet
- Naltrexon/Bupropion + Lifestyle (No Intervention): Naltrexon/Bupropion + Lifestyle

INTERVENTIONS:
Other: Very Low Calorie Diet — This is a parallel multicentric longitudinal randomized controlled trial in which prospective data will be collected from the electronic health record. The inclusion and exclusion criteria will be checked and afterwards patients will be randomized to (unblinded) medication only or combination with VLCKD. Both arms include NB and lifestyle changes for 26 weeks but the patients belonging to the experimental arm must follow a VLCKD in the first 10 weeks on top of it. Like the other arm, the remaining 16 weeks will consist of NB combined with lifestyle interventions. Afterwards there is a follow-up extension of 26 weeks.
  Arms: Naltrexon/Bupropion + Lifestyle + VLCKD

SUMMARY:
The goal of this clinical trial is to evaluate the superiority of combined VLCKD, intensive lifestyle intervention and naltrexone/bupropion (N/B) versus standard of care with naltrexone/bupropion on weight loss for people with weight regain after bariatric surgery.

The main questions it aims to answer are:

Primary endpoint:

• The percentage of weight loss at 26 weeks

Secondary endpoints:

* A weight loss percentage at 10 weeks, 16 weeks and at end of trial (= 52 weeks from start)
* A proportion of patients with a weight loss percentage of 5% or more at 10, 16, 26 and 52 weeks
* A proportion of patients with a weight loss percentage of 10% or more at 10, 16, 26 and 52 weeks
* The time to reach a weight loss percentage of 5% and 10%
* The dose of naltrexone/bupropion used at 10, 16, 26 and 52 weeks and at the end of the trial
* The tolerability of VLCKD and NB
* The adherence to VLCKD and NB
* The Patient-Reported Outcome Measures (PROMs) of hunger and cravings at 0, 4, 10, 16, 26 and 52 weeks
* The change in fasting glucose, lipids and blood pressure at 10, 16, 26 and 52 weeks

Researchers will compare an experimental arm (N/B + Lifestyle + VLCKD) with comparator arm (NB + lifestyle) to see if combined VLCKD, intensive lifestyle and N/B is superior.

Participants will:

* get NB and lifestyle changes for 26 weeks
* follow a VLCKD in the first 10 weeks on top of it, if they belong to the experimental arm
* follow NB combined with lifestyle the remaining 16 weeks
* be followed-up for an extension of 26 weeks
* come to the hospital at week 1, 10, 16, 26, 52

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for inclusion in this Trial must meet all of the following criteria:

  1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
  2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
  3. Miminum 18 years of age at the time of Informed Consent signature
  4. Underwent bariatric surgery (RYGB or SG) with weight regain ≥10% of nadir weight
  5. People without Type 2 diabetes (T2D) • No history, no drugs, HbA1c < 6,5% and FPG <126 mg/dl) All participants that are considered for Trial participation, per the above criteria will be documented on the Screening Log, including Screen Failures.

Exclusion Criteria:

* Participants eligible for this Trial must not meet any of the following criteria:

  1. Participant has a history of type 2 diabetes mellitus (also drugs, HbA1c > 6,5% and FPG >126 mg/dl)
  2. IFemale who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
  3. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
  4. Not willing to sign informed consent
  5. Younger than 18 years of age at the time of Informed Consent signature
  6. Other types of bariatric surgery other than RYGB or SG (including LAGB, BPD)
  7. Underwent bariatric surgery (RYGB or SG) with weight regain <10% of nadir weight
  8. Contraindication for VLCKD, including CKD stage 4-5, liver cirrhosis, type 1 diabetes mellitus, active gout
  9. Contraindication for NB including the use of opioids, history of CNS tumor or seizures, severe psychiatric disorder or > 2 psychotropic medications, uncontrolled hypertension
  10. Use of other drugs for weight management (e.g. GLP1Ra) in the last 3 months prior to trial intervention
  11. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol Participants who meet one or more of the above exclusion criteria must not proceed to be enrolled/randomized in the Trial and will be identified on the Screening Log as Screen Failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the superiority of combined VLCKD, intensive lifestyle intervention and naltrexone/bupropion versus standard of care with naltrexone/bupropion on weight loss. | 26 weeks
  The percentage of weight loss at 26 weeks

SECONDARY OUTCOMES:
• A weight loss percentage at 10 weeks, 16 weeks and at end of trial (= 52 weeks from start) | 10,16 and 52 weeks
  in %
• A proportion of patients with a weight loss percentage of 5% or more at 10, 16, 26 and 52 weeks | 10, 16, 26 and 52 weeks
  in %
• A proportion of patients with a weight loss percentage of 10% or more at 10, 16, 26 and 52 weeks | 10, 16, 26 and 52 weeks
  in %
• The time to reach a weight loss percentage of 5% and 10% | 52 weeks
  in weeks
• The dose of naltrexone/bupropion used at 10, 16, 26 and 52 weeks and at the end of the trial | 10, 16, 26 and 52 weeks
  the dose is in mg
• The tolerability of VLCKD | 52 weeks
  The amount of reported adverse effects, in relation to the achieved VLCKD.
• The tolerability of NB | 52 weeks
  The amount of reported adverse effects, in relation to the achieved dose level.
• The adherence to VLCKD | 52 weeks
  The amount meals eaten per day, in accordance to the dietary advice.
• The adherence to NB | 52 weeks
  The amount of tablets taken per day, in accordance with the medicinal advice.
• The change in fasting glucose at 10, 16, 26 and 52 weeks | at 10, 16, 26 and 52 weeks
  fasting glucose in mg/dl
• The change in lipids at 10, 16, 26 and 52 | at 10, 16, 26 and 52 weeks
  lipids in mg/dl
• The change in blood pressure at 10, 16, 26 and 52 | at 10, 16, 26 and 52 weeks
  blood pressure in mmHg

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge, Bruges, West-Vlaanderen

DOCUMENTS (1):
  • Study Protocol (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT06881485/Prot_000.pdf